CLINICAL TRIAL: NCT05469698
Title: Onsite Tobacco Cessation Treatment for Patients With Peripheral Artery Disease (PAD): A Feasibility Study
Brief Title: Onsite Tobacco Cessation Treatment for Patients With PAD
Acronym: PAD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12774
Record Dates: First submitted 2022-07-13; First posted 2022-07-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Tobacco Cessation; Peripheral Artery Disease
MeSH Terms: conditions — Tobacco Use Cessation; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard Care (Other): All participants will receive standard care by the Tobacco Treatment Research Program. This includes nicotine replacement therapy such as patches, gum, or lozenges, counseling by a Tobacco Treatment Specialist, and complete questionnaires.
  Interventions: Behavioral: Tobacco Treatment Research Program Standard Care

INTERVENTIONS:
Behavioral: Tobacco Treatment Research Program Standard Care — Participants interested in quitting tobacco will be offered standard tobacco cessation care including nicotine replacement therapy and counseling.

SUMMARY:
Tobacco cessation treatment is needed for individuals with peripheral artery disease (PAD) to improve symptoms, lower cardiovascular risk, and prevent amputation. While such treatment is effective, many PAD patients do not receive cessation therapy. Participants will receive nicotine replacement therapy, counseling, and and complete questionnaires. We hypothesize that integrating tobacco cessation services into a dedicated PAD clinic (OU CVI Limb Preservation Clinic) can improve tobacco cessation rates and improve PAD-related health outcomes in this at risk population.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosed peripheral artery disease
* Tobacco user
* 18 years of age or older
* Willing/able to attend all study visits
* Be able to read, speak, and understand English

Exclusion Criteria:

* Do not meet the specified inclusion criteria above

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Biochemically confirmed abstinence | 13 weeks post enrollment
  We will measure the biochemically-confirmed self-reported smoking cessation rate at 13 weeks post-enrollment (a cessation rate of ≥ 15-20% will be a sign of feasibility).

SECONDARY OUTCOMES:
Rate of enrollment | Duration of the study (approximately 6 months)
  We will measure the rate of enrollment over those approached to be in the study (≥ 25% enrolled will indicate feasibility).

OTHER OUTCOMES:
Improvements in PAD | Baseline to 13 weeks post enrollment
  We will evaluate improvements among participants based on their responses in surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Darla E Kendzor, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- TSET Health Promotion Research Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
: Yes De-identified data will be made available to investigators upon request, after publication of the primary study findings, and with a data-sharing agreement that specifies the investigator(s) will 1) use the data only for research purposes and not to identify any individual participant, 2) store the data on a secure device (e.g., encrypted, password-protected), and 3) destroy or return the data after completion of the analyses.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be made available to investigators upon request after publication of the primary study findings.
Access Criteria: Data sharing agreement